CLINICAL TRIAL: NCT04828161
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study of Ensovibep (MP0420) in Ambulatory Adult Patients With Symptomatic COVID-19 - The "EMPATHY" Trial
Brief Title: A Dose Finding, Efficacy and Safety Study of Ensovibep (MP0420) in Ambulatory Adult Patients With Symptomatic COVID-19
Acronym: EMPATHY
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Phase 2 completed as planned. Due to the evolving landscape of treatments for COVID-19, the placebo-controlled Phase 3 design will not proceed. No patients were actively participating at the time of termination.
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Molecular Partners AG (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP0420-CP302; 2021-000890-10 (EudraCT Number); CSKO136A12201J (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: COVID-19
Keywords: ensovibep; COVID-19 treatment, symptom reduction, viral load reduction,; EMPATHY; SARS-CoV-2; designed ankyrin repeat protein (DARPin®); angiotensin-converting enzyme 2 (ACE2)
MeSH Terms: conditions — COVID-19 | interventions — ensovibep

STUDY DESIGN:
Intervention Model Description: * Parallel: participants are assigned to one of two or more groups in parallel for the duration of the study.
  * 4 Arms under Phase 2 and 2 Arms under Phase 3
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * Double Blind: two or more parties are unaware of the intervention assignment
  * Masked roles are: Subject, Caregiver, Investigator or Outcomes Assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 2 / Part A, ensovibep active treatment arm 1 (Experimental): Phase 2 / Part A: ensovibep active treatment arm 1
  Interventions: Drug: ensovibep
- Phase 2 / Part A, ensovibep active treatment arm 2 (Experimental): Phase 2 / Part A: ensovibep active treatment arm 2
  Interventions: Drug: ensovibep
- Phase 2 / Part A, ensovibep active treatment arm 3 (Experimental): Phase 2 / Part A: ensovibep active treatment arm 3
  Interventions: Drug: ensovibep
- Phase 2 / Part A, Placebo (Placebo Comparator): Phase 2 / Part A: Placebo
  Interventions: Drug: Placebo
- Phase 3/ Part B, ensovibep active treatment arm 4 (Experimental): Phase 3/ Part B: ensovibep active treatment. Part B was not initiated.
  Interventions: Drug: ensovibep
- Phase 3/ Part B, Placebo arm (Placebo Comparator): Phase 3/ Part B: Placebo. Part B was not initiated.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ensovibep — IV on day 1 only.
  Other Names: MP0420
  Arms: Phase 2 / Part A, ensovibep active treatment arm 1; Phase 2 / Part A, ensovibep active treatment arm 2; Phase 2 / Part A, ensovibep active treatment arm 3; Phase 3/ Part B, ensovibep active treatment arm 4
Drug: Placebo — IV on day 1 only.
  Arms: Phase 2 / Part A, Placebo; Phase 3/ Part B, Placebo arm

SUMMARY:
The purpose of this study is to establish the antiviral efficacy of ensovibep against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in humans, identify the optimal dose, and demonstrate its clinical value for treating COVID-19 in adult ambulatory patients.

DETAILED DESCRIPTION:
Primary objectives:

Part A: The primary objective of this Part is to demonstrate superiority of ensovibep, compared to placebo, in reducing SARS-CoV-2 viral load through Day 8.

Part B: The primary objective of this Part is to demonstrate superiority of ensovibep, compared to placebo, in reducing the occurrence of hospitalizations (≥ 24 hours of acute care) and/or emergency room visits related to COVID-19 or death from any cause up to Day 29.

Secondary objectives:

Part A: The secondary objectives of this Part are:

* To assess the effect of ensovibep, compared to placebo, in reducing the occurrence of hospitalizations (≥ 24 hours of acute care) and/or emergency room visits related to COVID-19 or death from any cause up to Day 29
* To assess the effect of ensovibep, compared to placebo, in reducing COVID-19 symptoms through Day 29
* To evaluate safety and tolerability of ensovibep
* To characterize the pharmacokinetics (PK) of ensovibep

Part B: The secondary objectives of this Part are:

* To assess the effect of ensovibep, compared to placebo, in reducing SARS-CoV-2 viral load through Day 8
* To assess the effect of ensovibep, compared to placebo, in reducing COVID-19 symptoms up to Day 29
* To evaluate the immunogenicity of ensovibep during the study and its clinical relevance (PK, efficacy and safety)
* To evaluate safety and tolerability of ensovibep

Although Amendment 2 was created, modifications for this amendment are not reflected as it was never approved or implemented in the US. The study was conducted under Global Protocol Amendment 1, the last active version of the protocol.

ELIGIBILITY:
Part A Inclusion Criteria:

1. Men and women ≥ 18 years of age on the day of inclusion (no upper limit).
2. Presence of two or more of the following COVID-19 symptoms with an onset within 7 days of dosing: Feeling hot or feverish, cough, sore throat, low energy, or tiredness, headache, muscle or body aches, chills or shivering, and shortness of breath.
3. Positive test for SARS-CoV-2 in upper respiratory swab on the day of dosing (rapid antigen test).
4. Understand and agree to comply with the planned study procedures.
5. The patient or legally authorized representative give signed informed consent.

Part A Exclusion Criteria:

1. Requiring hospitalization at time of screening, or at time of study drug administration.
2. Oxygen saturation (SpO2) ≤ 93% on room air at sea level or ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2) < 300, respiratory rate ≥ 30 per minute, and heart rate ≥ 125 per minute. In India, patients with a respiratory rate ≥ 24 per minute or with an oxygen saturation ≤ 93% on room air (SpO2) are not eligible.
3. Known allergies to any of the components used in the formulation of the ensovibep or placebo.
4. Suspected or proven serious, active bacterial, fungal, viral, or other infection (besides SARS-CoV-2) that in the opinion of the investigator could constitute a risk when taking intervention.
5. Any serious concomitant systemic disease, condition, or disorder that, in the opinion of the investigator, should preclude participation in this study.
6. Any co-morbidity requiring surgery within 7 days of dosing, or that is considered life-threatening within 29 days of dosing.
7. Prior or concurrent use of any medication for treatment of COVID-19, including antiviral agents, convalescent serum, or anti-viral antibodies. Purely symptomatic therapies (e.g., over-the-counter [OTC] cough medications, acetaminophen, and nonsteroidal anti-inflammatory drugs [NSAIDs]) are permitted. Prior vaccination for COVID-19 is permitted.
8. Are concurrently enrolled or were enrolled within the last 30 days or within 5 half-lives (whichever is longer) in any other type of medical research judged not to be scientifically or medically compatible with this study.
9. Are pregnant or breast feeding.
10. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception at the time of dosing and for 11 weeks after dosing of study drug. Highly effective contraception methods include:

    1. Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (i.e., calendar, ovulation, symptothermal, and postovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Female sterilization (have had bilateral surgical oophorectomy [with or without hysterectomy], total hysterectomy, or bilateral tubal ligation at least 6 weeks before taking study treatment). In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
    3. Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that patient.
    4. Use of oral, injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment. If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the informed consent form (ICF).
11. Patients in the USA who are at high risk of progression to severe COVID-19 illness or hospitalization must not be enrolled in Part A of this study as a placebo-controlled study may not be appropriate in this patient population due to the availability of anti-viral mAbs under EUA in the USA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (27):
  - Jasper Summit Research, LLC, Jasper, Alabama
  - Benchmark Southern California, Colton, California
  - Ascada Research, Fullerton, California
  - Pacific Neuropsychiatric Specialists, Mission Viejo, California
  - Providence Family Medical Center, Redondo Beach, California
  - Future Innovative Treatments, Colorado Springs, Colorado
  - Boward Infectious Disease and Primary Care, Margate, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Life Spring Research Foundation, Miami, Florida
  - Bio-Medical Research, LLC, Miami, Florida
  - Panax Clinical Research, LLC, Miami Lakes, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Gwinnett Research Institute, Buford, Georgia
  - IACT Health, Columbus, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Centennial Medical Group - Research Department, Elkridge, Maryland
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Monroe Biomedical Research, Monroe, North Carolina
  - Wilmington Health, Wilmington, North Carolina
  - VitaLink Research, Greenville, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Fairway Medical Clinic, Houston, Texas
  - 1960 Family Practice, PA, Houston, Texas
  - Zion Urgent Care Clinic, Katy, Texas
  - Family Practice Center, McAllen, Texas
  - Epic Medical Research, Red Oak, Texas
- Debreceni Egyetem, Debrecen, Hungary
- India (10):
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - BAPS Pramukhswami Hospital, Surat, Gujarat
  - Durgabai Deshmukh Hospital & Research Centre, Vidyānagar, Hyderabad
  - Shetty's Hospital, Bengaluru, Karnataka
  - Government Medical College, Aurangabad, Maharashtra
  - Grant Medical College & Sir J. J. Group of Hospitals, Mumbai, Maharashtra
  - Government Medical College and Hospital, Nagpur, Maharashtra
  - All India Institute of Medical Sciences - Nagpur, Nagpur, Maharashtra
  - VHS-Infectious Disease Medical Centre, Chennai, Tamil Nadu
  - St. Theresa's Hospital, Hyderabad, Telangana
- UMC Utrecht, Utrecht, Netherlands
- South Africa (9):
  - FARMOVS (Pty) Ltd, Bloemfontein, Free State
  - Sandton Medical Research Centre, Sandton, Gauteng
  - George Provincial Hospital, George, Western Cape
  - Dr JM Engelbrecht Trial Site, Somerset West, Western Cape
  - Enhancing Care Foundation, Durban
  - Clinresco Centres (Pty) Ltd, Kempton Park
  - DJW Navorsing, Krugersdorp
  - Jongaie Research, Pretoria
  - Wits Clinical Research, Soweto

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1428

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 2 parts, Part A and Part B. The Part A was Phase II proof of efficacy study conducted in ambulatory adult participants with symptomatic coronavirus disease 2019 (COVID-19) at 45 centers across 5 countries (Hungary, India, Netherlands, South Africa, and USA) between 10 May 2021 and 27 Jan 2022. The Part B was to be a Phase III confirmatory study. Only Part A analysis is reported since Part B of the study was not initiated.
Pre-assignment Details: The Part A of the study consisted of a screening period (up to 3 days) followed by study treatment on Day 1. Participants were randomized in 1:1:1:1 ratio, stratified by risk for COVID-19 disease progression, to receive 1 of 4 study treatments (Ensovibep 600 mg or Ensovibep 225 mg or Ensovibep 75 mg or Placebo). A total of 407 participants were randomized in the study, of which 400 were treated.
Groups:
- Ensovibep 600 mg: Participants received single intravenous (IV) infusion of ensovibep 600 milligram (mg) on Day 1.
- Ensovibep 225 mg: Participants received single IV infusion of ensovibep 225 mg on Day 1.
- Ensovibep 75 mg: Participants received single IV infusion of ensovibep 75 mg on Day 1.
- Placebo: Participants received single IV infusion of placebo matching with ensovibep on Day 1.
Period: Overall Study
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg | Placebo
Started (Randomized) | 100 | 102 | 103 | 102
Completed | 97 | 95 | 96 | 94
Not Completed | 3 | 7 | 7 | 8
Not completed — Withdrawal by Subject | 0 | 3 | 3 | 4
Not completed — Lost to Follow-up | 1 | 4 | 2 | 2
Not completed — Other | 2 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants in the randomized set for whom IV infusion of study treatment was initiated during the treatment period.
Groups:
- Ensovibep 600 mg: Participants received single IV infusion of ensovibep 600 mg on Day 1.
- Total: Total of all reporting groups
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg | Placebo | Total
Number analyzed (Participants) | 100 | 100 | 101 | 99 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (11.50) | 40.2 (12.90) | 41.5 (12.84) | 42.3 (13.75) | 41.1 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 54 | 60 | 57 | 218
  Male | 53 | 46 | 41 | 42 | 182
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 59 | 63 | 62 | 63 | 247
  Asian | 14 | 14 | 13 | 16 | 57
  Black or African American | 16 | 11 | 14 | 11 | 52
  Multiple | 5 | 4 | 6 | 8 | 23
  Not reported | 1 | 4 | 3 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2 | 0 | 4
  American Indian or Alaska Native | 3 | 0 | 1 | 0 | 4
  Unknown | 1 | 3 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part A: Time-Weighted Change From Baseline in Log10 Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Viral Load Through Day 8
Description: The SARS-CoV-2 viral load was measured by means of a nasopharyngeal swab, followed by quantitative reverse transcription-polymerase chain reaction assay at a central laboratory. The multiple comparison procedure-modeling methodology was used. Time-weighted change from baseline was used as viral loads were measured at multiple time points.
Time Frame: Baseline (Day 1) and Days 3, 5 and 8
Population: The FAS included all participants in the randomized set for whom IV infusion of study treatment was administered. Only participants included in the analysis are reported.
Measure: Least Squares Mean (Standard Error); unit: log10 copies/milliliter (mL)
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg | Placebo
Number analyzed (Participants) | 89 | 97 | 97 | 87
log10 copies/milliliter (mL) | -1.99 (0.097) | -1.73 (0.093) | -1.81 (0.093) | -1.40 (0.098)
Statistical Analysis 1: Comparison: Ensovibep 600 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Least square (LS) mean difference = -0.59, 95% CI 2-sided [-0.86 to -0.32], Standard Error of Mean 0.138
Statistical Analysis 2: Comparison: Ensovibep 225 mg vs Placebo; Test type: Superiority; p = 0.014, ANCOVA; LS mean difference = -0.33, 95% CI 2-sided [-0.60 to -0.07], Standard Error of Mean 0.135
Statistical Analysis 3: Comparison: Ensovibep 75 mg vs Placebo; Test type: Superiority; p = 0.002, ANCOVA; LS mean difference = -0.42, 95% CI 2-sided [-0.68 to -0.15], Standard Error of Mean 0.135

2. Secondary Outcome: Part A: Percentage of Participants With Hospitalizations and/or ER Visits Related to COVID-19 or Death From Any Cause
Description: Percentage of participants experiencing hospitalizations (>= 24 h of acute care) and/or ER visits related to COVID-19 or death from any cause up to Day 29 were presented along with relative risk to placebo.
Time Frame: Up to Day 29
Population: The FAS included all participants in the randomized set for whom IV infusion of study treatment was administered.
Measure: Number; unit: percentage of participants
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg | Placebo
Number analyzed (Participants) | 100 | 100 | 101 | 99
percentage of participants
  Any event | 1.0 | 3.0 | 0.0 | 6.1
  Hospitalizations (≥ 24 h of acute care) | 0.0 | 2.0 | 0.0 | 5.1
  Emergency room visits related to COVID-19 | 1.0 | 1.0 | 0.0 | 5.1
  Death from any cause | 0.0 | 0.0 | 0.0 | 2.0

3. Secondary Outcome: Part A: Time to Sustained Clinical Recovery
Description: Sustained clinical recovery was defined as follows;
  1. All symptoms from the modified Food and Drug Administration (FDA) COVID-19 questionnaire scored as moderate or severe at baseline were subsequently scored as mild or absent, and
  2. All symptoms from the modified FDA COVID-19 questionnaire scored as mild or absent at baseline were subsequently scored as absent, with no subsequent worsening, up to Day 29.
Time Frame: Up to Day 29
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg | Placebo
Number analyzed (Participants) | 63 | 66 | 74 | 70
days | 23.0 [14.0 to 29.0] | 15.0 [13.0 to 21.0] | 14.0 [11.0 to 28.0] | 29.0 [21.0 to 32.0]

4. Secondary Outcome: Part A: Observed Maximum Serum Concentration (Cmax) of Total and Free Ensovibep
Description: Blood samples were collected to determine the Cmax of free ensovibep (ensovibep not bound to target) and total ensovibep (sum of ensovibep not bound to and bound to target) concentrations in serum.
Time Frame: Data was summarized from pre-dose and at 15 minutes and 90 minutes after end of study drug infusion on Day 1, and at Days 3, 8, 15, 29, 61 and 91
Population: The Pharmacokinetic (PK) analysis set included all participants with at least 1 available valid (that is, not flagged for exclusion) PK concentration measurement, who received any study treatment and with no protocol deviations that impacted PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (mcg) per mL
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg
Number analyzed (Participants) | 94 | 92 | 95
microgram (mcg) per mL
  Total Ensovibep: number analyzed (Participants) | 94 | 90 | 93
  Total Ensovibep | 187 (25.3) | 70.4 (27.5) | 25.1 (38.4)
  Free Ensovibep | 210 (26.3) | 78.1 (31.5) | 29.3 (46.4)

5. Secondary Outcome: Part A: Area Under the Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Total and Free Ensovibep
Description: Blood samples were collected to determine the AUClast of free ensovibep (ensovibep not bound to target) and total ensovibep (sum of ensovibep not bound to and bound to target) concentrations in serum.
Time Frame: as for outcome 4
Population: The PK analysis set included all participants with at least 1 available valid (that is, not flagged for exclusion) PK concentration measurement, who received any study treatment and with no protocol deviations that impacted PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg
Number analyzed (Participants) | 94 | 91 | 95
h*mcg/mL
  Total Ensovibep: number analyzed (Participants) | 94 | 88 | 95
  Total Ensovibep | 63300 (87.6) | 21100 (122.0) | 7950 (67.1)
  Free Ensovibep | 68200 (84.4) | 22500 (126.9) | 8380 (67.9)

6. Secondary Outcome: Part A: Area Under the Concentration-Time Curve From Time Zero to 48 Hours (AUC 0-48h) of Total and Free Ensovibep
Description: Blood samples were collected to determine the AUC 0-48h of free ensovibep (ensovibep not bound to target) and total ensovibep (sum of ensovibep not bound to and bound to target) concentrations in serum.
Time Frame: Data was summarized from pre-dose and at 15 minutes and 90 minutes after end of study drug infusion on Day 1, and at Day 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg
Number analyzed (Participants) | 95 | 90 | 95
h*mcg/mL
  Total Ensovibep: number analyzed (Participants) | 93 | 89 | 95
  Total Ensovibep | 7520 (35.3) | 2830 (35.7) | 999 (34.4)
  Free Ensovibep | 8290 (32.1) | 2800 (156.2) | 1120 (36.7)

7. Secondary Outcome: Part A: Area Under the Concentration-Time Curve From Time Zero to 168 Hours (AUC 0-168h) of Total and Free Ensovibep
Description: Blood samples were collected to determine the AUC 0-168h of free ensovibep (ensovibep not bound to target) and total ensovibep (sum of ensovibep not bound to and bound to target) concentrations in serum.
Time Frame: Data was summarized from pre-dose and at 15 minutes and 90 minutes after end of study drug infusion on Day 1, and at Days 3 and 8
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg
Number analyzed (Participants) | 95 | 89 | 95
h*mcg/mL
  Total Ensovibep: number analyzed (Participants) | 93 | 89 | 94
  Total Ensovibep | 23000 (23.7) | 8570 (33.1) | 3020 (31.4)
  Free Ensovibep | 25200 (23.2) | 8940 (73.2) | 3390 (35.3)

8. Secondary Outcome: Part A: Area Under the Concentration-Time Curve From Time Zero to 336 Hours (AUC 0-336h) of Total and Free Ensovibep
Description: Blood samples were collected to determine the AUC 0-336h of free ensovibep (ensovibep not bound to target) and total ensovibep (sum of ensovibep not bound to and bound to target) concentrations in serum.
Time Frame: Data was summarized from pre-dose and at 15 minutes and 90 minutes after end of study drug infusion on Day 1, and at Days 3, 8 and 15
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg
Number analyzed (Participants) | 95 | 88 | 94
h*mcg/mL
  Total Ensovibep: number analyzed (Participants) | 93 | 87 | 93
  Total Ensovibep | 38200 (23.2) | 13800 (37.6) | 5040 (31.9)
  Free Ensovibep | 41800 (23.5) | 15300 (41.6) | 5620 (39.1)

9. Secondary Outcome: Part A: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUCinfinity) of Total and Free Ensovibep
Description: Blood samples were collected to determine the AUCinfinity of free ensovibep (ensovibep not bound to target) and total ensovibep (sum of ensovibep not bound to and bound to target) concentrations in serum.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg
Number analyzed (Participants) | 87 | 82 | 82
h*mcg/mL
  Total Ensovibep: number analyzed (Participants) | 87 | 77 | 82
  Total Ensovibep | 75400 (33.5) | 27600 (36.3) | 9930 (41.0)
  Free Ensovibep: number analyzed (Participants) | 87 | 82 | 80
  Free Ensovibep | 80100 (40.6) | 29400 (34.8) | 9540 (45.8)

10. Secondary Outcome: Part A: Time to Reach the Maximum Concentration (Tmax) of Total and Free Ensovibep
Description: Blood samples were collected to determine the Tmax of free ensovibep (ensovibep not bound to target) and total ensovibep (sum of ensovibep not bound to and bound to target) concentrations in serum.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg
Number analyzed (Participants) | 95 | 92 | 95
hour
  Total Ensovibep: number analyzed (Participants) | 95 | 90 | 92
  Total Ensovibep | 0.935 (457.5) | 1.30 (693.5) | 1.05 (573.6)
  Free Ensovibep | 1.01 (473.8) | 1.09 (516.6) | 1.24 (810.1)

11. Secondary Outcome: Part A: Apparent Total Body Clearance (CL) of Total and Free Ensovibep
Description: Blood samples were collected to determine the CL of free ensovibep (ensovibep not bound to target) and total ensovibep (sum of ensovibep not bound to and bound to target) concentrations in serum.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg
Number analyzed (Participants) | 84 | 80 | 74
mL/h
  Total Ensovibep: number analyzed (Participants) | 77 | 78 | 74
  Total Ensovibep | 8.07 (35.4) | 8.11 (36.1) | 7.48 (42.1)
  Free Ensovibep | 7.55 (37.3) | 7.64 (35.3) | 7.78 (43.0)

12. Secondary Outcome: Part A: Terminal Elimination Rate Constant (Lambda z) of Total and Free Ensovibep
Description: Blood samples were collected to determine the lambda z of free ensovibep (ensovibep not bound to target) and total ensovibep (sum of ensovibep not bound to and bound to target) concentrations in serum.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg
Number analyzed (Participants) | 84 | 79 | 74
per hour
  Total Ensovibep: number analyzed (Participants) | 83 | 70 | 72
  Total Ensovibep | 0.003 (52.1) | 0.002 (50.6) | 0.002 (39.5)
  Free Ensovibep | 0.003 (69.6) | 0.003 (48.3) | 0.003 (61.2)

13. Secondary Outcome: Part A: Terminal Elimination Half-Life (T1/2) of Total and Free Ensovibep
Description: Blood samples were collected to determine the T1/2 of free ensovibep (ensovibep not bound to target) and total ensovibep (sum of ensovibep not bound to and bound to target) concentrations in serum.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg
Number analyzed (Participants) | 90 | 83 | 83
hour
  Total Ensovibep: number analyzed (Participants) | 89 | 81 | 83
  Total Ensovibep | 274 (54.0) | 290 (53.8) | 309 (39.8)
  Free Ensovibep: number analyzed (Participants) | 90 | 83 | 81
  Free Ensovibep | 262 (67.7) | 234 (48.3) | 215 (60.6)

14. Secondary Outcome: Part A: Apparent Volume of Distribution (Vz) of Total and Free Ensovibep
Description: Blood samples were collected to determine the Vz of free ensovibep (ensovibep not bound to target) and total ensovibep (sum of ensovibep not bound to and bound to target) concentrations in serum.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg
Number analyzed (Participants) | 84 | 80 | 74
mL
  Total Ensovibep: number analyzed (Participants) | 77 | 78 | 74
  Total Ensovibep | 3230 (35.0) | 3310 (37.5) | 3330 (38.7)
  Free Ensovibep | 2760 (46.1) | 2590 (36.4) | 2470 (45.6)

15. Primary Outcome: Part B: Percentage of Participants With Hospitalizations and/or Emergency Room (ER) Visits Related to COVID-19 or Death From Any Cause
Description: Percentage of participants experiencing hospitalizations [>= 24 hour (h) of acute care] and/or ER visits related to COVID-19 or death from any cause up to Day 29.
Time Frame: Up to Day 29
Population: The Part B of the study was not initiated based on regulatory feedback indicating that with evolving treatment options, a placebo controlled design was no longer considered to be appropriate.
Groups:
- Phase 3/Part B: Ensovibep 75 mg: Phase 3/Part B: ensovibep active treatment. Part B was not initiated.
- Phase 3/Part B: Placebo: Phase 3/Part B: Placebo. Part B was not initiated.
Arm/Group | Phase 3/Part B: Ensovibep 75 mg | Phase 3/Part B: Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Part B: Change From Baseline in Log10 SARS-CoV-2 Viral Load Through Day 8
Description: The SARS-CoV-2 viral load was measured by means of a nasopharyngeal swab, followed by quantitative reverse transcription-polymerase chain reaction assay at a central laboratory. The multiple comparison procedure-modeling methodology was used.
Time Frame: Baseline (Day 1) and Days 3, 5 and 8
Population: as for outcome 15
Arm/Group | Phase 3/Part B: Ensovibep 75 mg | Phase 3/Part B: Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Part B: Time to Sustained Clinical Recovery
Description: Sustained clinical recovery was defined as follows;
  1. All symptoms from the modified FDA COVID-19 questionnaire scored as moderate or severe at baseline were subsequently scored as mild or absent, and
  2. All symptoms from the modified FDA COVID-19 questionnaire scored as mild or absent at baseline were subsequently scored as absent, with no subsequent worsening, up to Day 29.
Time Frame: Up to Day 29
Population: as for outcome 15
Arm/Group | Phase 3/Part B: Ensovibep 75 mg | Phase 3/Part B: Placebo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Part B: Percentage of Participants With Treatment-Emergent Anti-Drug Antibody (ADA) Response to Ensovibep
Description: Treatment-emergent ADA is defined as any participant with a
  1. 2-fold (1 dilution) increase in titer than the minimum required dilution if no ADAs were detected at baseline (treatment-induced ADA); or,
  2. 4-fold (2 dilutions) increase in titer compared with baseline if ADAs were detected at baseline (treatment-boosted ADA).
Time Frame: Pre-dose on Day 1 and Days 15, 29, 61 and 91 postdose of Ensovibep
Population: as for outcome 15
Arm/Group | Phase 3/Part B: Ensovibep 75 mg | Phase 3/Part B: Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were reported from first dose of study treatment (Day 1) until end of study treatment, up to a maximum duration of 98 days.
Groups:
- Ensovibep Total: Participants received single IV infusion of ensovibep on Day 1.
Arm/Group | Ensovibep 600 mg | Ensovibep 225 mg | Ensovibep 75 mg | Ensovibep Total | Placebo
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/98 | 0/102 | 0/300 | 2/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 2/98 | 1/102 | 3/300 | 9/100
Other Adverse Events (participants affected / at risk) | 51/100 | 40/98 | 40/102 | 131/300 | 53/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ensovibep 600 mg (N=100) | Ensovibep 225 mg (N=98) | Ensovibep 75 mg (N=102) | Ensovibep Total (N=300) | Placebo (N=100)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cor pulmonale (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 4
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ensovibep 600 mg (N=100) | Ensovibep 225 mg (N=98) | Ensovibep 75 mg (N=102) | Ensovibep Total (N=300) | Placebo (N=100)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 3 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 4 | 8 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 1
Disorder of globe (Eye disorders) | 0 | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 1 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 4 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1 | 6 | 1
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 1 | 3 | 1
Infusion site haematoma (General disorders) | 0 | 0 | 0 | 0 | 2
Infusion site swelling (General disorders) | 0 | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 1 | 3 | 0
Pain (General disorders) | 1 | 1 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Swelling face (General disorders) | 0 | 0 | 1 | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 1 | 2 | 0
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0
Allergy to chemicals (Immune system disorders) | 0 | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
COVID-19 (Infections and infestations) | 6 | 2 | 1 | 9 | 4
COVID-19 pneumonia (Infections and infestations) | 2 | 2 | 0 | 4 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Eye infection bacterial (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Genital infection fungal (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 1 | 3 | 9 | 5
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Pancreatitis viral (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 2 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 3 | 1 | 1 | 5 | 1
Alanine aminotransferase increased (Investigations) | 7 | 3 | 1 | 11 | 2
Amylase increased (Investigations) | 4 | 1 | 1 | 6 | 2
Aspartate aminotransferase increased (Investigations) | 6 | 3 | 1 | 10 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 3 | 0 | 1 | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 1 | 1 | 5 | 1
Blood creatinine increased (Investigations) | 6 | 4 | 3 | 13 | 6
Blood glucose increased (Investigations) | 1 | 0 | 1 | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 2 | 0 | 0 | 2 | 1
Blood pressure increased (Investigations) | 0 | 1 | 1 | 2 | 1
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 1 | 1
Blood sodium increased (Investigations) | 0 | 0 | 1 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 3 | 1 | 4 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 1 | 2 | 0
Fibrin D dimer increased (Investigations) | 5 | 2 | 4 | 11 | 3
Gamma-glutamyltransferase increased (Investigations) | 3 | 1 | 3 | 7 | 1
Haematocrit decreased (Investigations) | 0 | 1 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 2 | 0 | 0 | 2 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 2
Lipase increased (Investigations) | 6 | 0 | 3 | 9 | 1
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1
Monocyte count decreased (Investigations) | 0 | 0 | 1 | 1 | 1
Monocyte count increased (Investigations) | 0 | 0 | 1 | 1 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 1 | 0 | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 3
Serum ferritin decreased (Investigations) | 0 | 0 | 1 | 1 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 2 | 4 | 8 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 1 | 3 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 4 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 2 | 5 | 0
Phlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Part B was not initiated based on regulatory feedback indicating that with evolving treatment options, a placebo controlled design was no longer considered to be appropriate. 2 patients randomized to ensovibep 225 mg didn't receive treatment they were randomized to: 1 patient received no active drug as infusion was not prepared correctly; 1 patient received lower dose (<75 mg) as infusion was interrupted. For Safety set, these 2 were reported in placebo and ensovibep 75 mg arms, respectively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT04828161/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT04828161/SAP_001.pdf